CLINICAL TRIAL: NCT05310162
Title: Effect of the Intervention "Food, Fun and Family" on Sleep Bruxism in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Claudia Cecilia Restrepo Serna, CES-LPH research group director, CES University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1017
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Sleep Bruxism, Childhood
Keywords: Children; Sleep bruxism; Added sugar; Screen time
MeSH Terms: conditions — Sleep Bruxism | interventions — Food; Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food, fun and family (Experimental): This intervention aims to change eating and screen time habits in children to decrease the amount of added sugar consumed and the time spent using recreational screens, this with guides and precise instructions given to the parents to have a healthier lifestyle.
  Interventions: Behavioral: Food, fun and family
- Counseling (Active Comparator): The parents will receive simple verbal instructions to reduce the consumption of added sugar and recreational screen time, giving advice on which foods to avoid and the amount of time permitted for the use of screens.
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Food, fun and family — The intervention consists of a series of change of habits in the way children eat, the reduction of the recreational time of screens and healthy habits of physical activity. This intervention, which is called "Food, Fun & Family (FFF)", is aimed at parents and has been shown to be effective in reducing the consumption of "empty calories" by children. It teaches parents skills to reduce their daily energy intake of added sugars and saturated fats, it also seeks to reduce screen time.
  The intervention contains information and recommendations, through guides, in which precise instructions are given about how to maintain a healthy environment at home.
  Other Names: FFF
  Arms: Food, fun and family
Behavioral: Counseling — Simple verbal instructions will be given in the consultation to reduce the time of use of screens and refined sugar.
  For refined sugar reduction, parents will be told to avoid sugary drinks, add sugar to drinks (juices, milk, etc.), and avoid snacks and sweets. It will also be indicated that the screen time should be less than two hours a day and in no case use them two hours before sleeping.
  Arms: Counseling

SUMMARY:
Excess consumption of refined sugar and increased use of recreational screen time are risk factors for alterations in the quality of life that have been associated with sleep bruxism in children and that compromise the same mechanisms of alteration of the reward system in the brain. Therefore, the question of this research is: What is the effect of the Intervention "Food, Fun and Family (FFF)" on the frequency of sleep bruxism in children? The general objective of the research is to evaluate the effect of the Intervention "Food, Fun and Family (FFF)" on the frequency of sleep bruxism in 84 children who attend the pediatric dentistry postgraduate clinic of the CES University and the private consultation Dr. Claudia Restrepo and Dr. Adriana Santamaría. The frequency of sleep bruxism will be evaluated with the translated and validated Spanish version of the Children's Sleep Habits Questionnaire (CSHQ), which will be answered by the parents. The consumption of added sugar will be evaluated with the version translated into Spanish of the Health Behavior in School-Aged Children - Food-Frequency Questionnaire (HBSC-FFQ). The time on screens will be recorded through the parents' report, of the time in hours that the child spends using electronic media in a recreational way each weekday for a week and each weekend day for a week.

A decrease in the frequency of sleep bruxism is expected to be found by reducing sugar consumption and screen time in the children evaluated.

The results of this study will be presented at the IADR, ACFO, ACOP and CES University research meetings and will be published in a peer-reviewed scientific journal in category Q1.

ELIGIBILITY:
Inclusion Criteria:

* Children who eat breakfast, lunch and dinner at home.
* Children whose feeding and habits management (upbringing) is in charge of the same group of representative adults.
* Children who live with their parents.
* Children attending the consultation for the first time.

Exclusion Criteria:

* Symptoms of respiratory disorders reported by parents in the CSHQ.
* Food allergies.
* Special diet restrictions.
* Developmental disorder influencing diet or weight.
* Basic endocrinological diseases.
* Being under endocrinological treatment.
* Previously diagnosed sleep disorders.
* Children who miss more than two assigned appointments.
* Parents of children who withdraw informed consent.
* Children who are diagnosed during the study with respiratory disorders.
* Children who are diagnosed during the study with food allergies.
* Children who for personal reasons cannot continue in the study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-04-11 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-05-05 (Estimated)

PRIMARY OUTCOMES:
Frecuency of sleep bruxism | 8 weeks
  Report from the parents in the CSHQ with values of usually, some times and no/rarely

SECONDARY OUTCOMES:
Frecuency of added sugar consumption | 8 weeks
  Report from the parents with the Spanish translated version of the HBSC-FFQ with values of never, less than one time a week, once a week, four days a week, five to six times a week, once a day every day, more than one a day
Screen time | 8 weeks
  Report from the parents of time in hours spent in front of audiovisuals, every day of the week during a week and each day of the weekend during a weekend

CONTACTS AND LOCATIONS:
Overall Officials: Claudia C Restrepo, PHD, Principal Investigator — CES LPH research group; Ruben D Manrique, PHD, Study Chair — CES LPH research group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lobbezoo F, Ahlberg J, Raphael KG, Wetselaar P, Glaros AG, Kato T, Santiago V, Winocur E, De Laat A, De Leeuw R, Koyano K, Lavigne GJ, Svensson P, Manfredini D. International consensus on the assessment of bruxism: Report of a work in progress. J Oral Rehabil. 2018 Nov;45(11):837-844. doi: 10.1111/joor.12663. Epub 2018 Jun 21. PMID 29926505
- [Background] Manfredini D, Restrepo C, Diaz-Serrano K, Winocur E, Lobbezoo F. Prevalence of sleep bruxism in children: a systematic review of the literature. J Oral Rehabil. 2013 Aug;40(8):631-42. doi: 10.1111/joor.12069. Epub 2013 May 24. PMID 23700983
- [Background] Fisberg M, Kovalskys I, Gomez G, Rigotti A, Sanabria LYC, Garcia MCY, Torres RGP, Herrera-Cuenca M, Zimberg IZ, Koletzko B, Pratt M, Aznar LAM, Guajardo V, Fisberg RM, Sales CH, Previdelli AN; ELANS Study Group. Total and Added Sugar Intake: Assessment in Eight Latin American Countries. Nutrients. 2018 Mar 22;10(4):389. doi: 10.3390/nu10040389. PMID 29565308
- [Background] Wittekind A, Walton J. Worldwide trends in dietary sugars intake. Nutr Res Rev. 2014 Dec;27(2):330-45. doi: 10.1017/S0954422414000237. PMID 25623085
- [Background] Newens KJ, Walton J. A review of sugar consumption from nationally representative dietary surveys across the world. J Hum Nutr Diet. 2016 Apr;29(2):225-40. doi: 10.1111/jhn.12338. Epub 2015 Oct 10. PMID 26453428
- [Background] Ervin RB, Kit BK, Carroll MD, Ogden CL. Consumption of added sugar among U.S. children and adolescents, 2005-2008. NCHS Data Brief. 2012 Mar;(87):1-8. PMID 22617043
- [Background] Lissak G. Adverse physiological and psychological effects of screen time on children and adolescents: Literature review and case study. Environ Res. 2018 Jul;164:149-157. doi: 10.1016/j.envres.2018.01.015. Epub 2018 Feb 27. PMID 29499467
- [Background] Ramos-Lopez O, Panduro A, Rivera-Iniguez I, Roman S. Dopamine D2 receptor polymorphism (C957T) is associated with sugar consumption and triglyceride levels in West Mexicans. Physiol Behav. 2018 Oct 1;194:532-537. doi: 10.1016/j.physbeh.2018.07.004. Epub 2018 Jul 4. PMID 30008437
- [Background] Yen JY, Ko CH, Yen CF, Wu HY, Yang MJ. The comorbid psychiatric symptoms of Internet addiction: attention deficit and hyperactivity disorder (ADHD), depression, social phobia, and hostility. J Adolesc Health. 2007 Jul;41(1):93-8. doi: 10.1016/j.jadohealth.2007.02.002. Epub 2007 Apr 12. PMID 17577539
- [Background] Del-Ponte B, Quinte GC, Cruz S, Grellert M, Santos IS. Dietary patterns and attention deficit/hyperactivity disorder (ADHD): A systematic review and meta-analysis. J Affect Disord. 2019 Jun 1;252:160-173. doi: 10.1016/j.jad.2019.04.061. Epub 2019 Apr 10. PMID 30986731
- [Background] Restrepo C, Manfredini D, Lobbezoo F. Sleep behaviors in children with different frequencies of parental-reported sleep bruxism. J Dent. 2017 Nov;66:83-90. doi: 10.1016/j.jdent.2017.08.005. Epub 2017 Aug 12. PMID 28807776
- [Background] Bach SL, Moreira FP, Goettems ML, Brancher LC, Oses JP, da Silva RA, Jansen K. Salivary cortisol levels and biological rhythm in schoolchildren with sleep bruxism. Sleep Med. 2019 Feb;54:48-52. doi: 10.1016/j.sleep.2018.09.031. Epub 2018 Oct 28. PMID 30529777
- [Background] Velez AL, Restrepo CC, Pelaez-Vargas A, Gallego GJ, Alvarez E, Tamayo V, Tamayo M. Head posture and dental wear evaluation of bruxist children with primary teeth. J Oral Rehabil. 2007 Sep;34(9):663-70. doi: 10.1111/j.1365-2842.2007.01742.x. PMID 17716265
- [Background] Souto-Souza D, Mourao PS, Barroso HH, Douglas-de-Oliveira DW, Ramos-Jorge ML, Falci SGM, Galvao EL. Is there an association between attention deficit hyperactivity disorder in children and adolescents and the occurrence of bruxism? A systematic review and meta-analysis. Sleep Med Rev. 2020 Oct;53:101330. doi: 10.1016/j.smrv.2020.101330. Epub 2020 May 19. PMID 32554210
- [Background] Turkoglu S, Akca OF, Turkoglu G, Akca M. Psychiatric disorders and symptoms in children and adolescents with sleep bruxism. Sleep Breath. 2014 Sep;18(3):649-54. doi: 10.1007/s11325-013-0928-y. Epub 2013 Dec 28. PMID 24371001
- [Background] Restrepo C, Santamaria A, Manrique R. Sleep bruxism in children: relationship with screen-time and sugar consumption. Sleep Med X. 2021 Apr 24;3:100035. doi: 10.1016/j.sleepx.2021.100035. eCollection 2021 Dec. PMID 34169271
- [Background] Manfredini D, Lobbezoo F, Giancristofaro RA, Restrepo C. Association between proxy-reported sleep bruxism and quality of life aspects in Colombian children of different social layers. Clin Oral Investig. 2017 May;21(4):1351-1358. doi: 10.1007/s00784-016-1901-5. Epub 2016 Jul 14. PMID 27417100
- [Background] Scariot R, Brunet L, Olsson B, Palinkas M, Regalo SCH, Rebellato NLB, Brancher JA, Torres CP, Diaz-Serrano KV, Kuchler EC, Zielak JC. Single nucleotide polymorphisms in dopamine receptor D2 are associated with bruxism and its circadian phenotypes in children. Cranio. 2022 Mar;40(2):152-159. doi: 10.1080/08869634.2019.1705629. Epub 2019 Dec 23. PMID 31868570
- [Background] Shqair AQ, Pauli LA, Costa VPP, Cenci M, Goettems ML. Screen time, dietary patterns and intake of potentially cariogenic food in children: A systematic review. J Dent. 2019 Jul;86:17-26. doi: 10.1016/j.jdent.2019.06.004. Epub 2019 Jun 19. PMID 31228564
- [Background] Lavigne GJ, Kato T, Kolta A, Sessle BJ. Neurobiological mechanisms involved in sleep bruxism. Crit Rev Oral Biol Med. 2003;14(1):30-46. doi: 10.1177/154411130301400104. PMID 12764018
- [Background] Horowitz-Kraus T, Hutton JS. Brain connectivity in children is increased by the time they spend reading books and decreased by the length of exposure to screen-based media. Acta Paediatr. 2018 Apr;107(4):685-693. doi: 10.1111/apa.14176. Epub 2017 Dec 27. PMID 29215151
- [Background] Cohen JFW, Rifas-Shiman SL, Young J, Oken E. Associations of Prenatal and Child Sugar Intake With Child Cognition. Am J Prev Med. 2018 Jun;54(6):727-735. doi: 10.1016/j.amepre.2018.02.020. Epub 2018 Apr 16. PMID 29674185
- [Background] Twenge JM, Campbell WK. Associations between screen time and lower psychological well-being among children and adolescents: Evidence from a population-based study. Prev Med Rep. 2018 Oct 18;12:271-283. doi: 10.1016/j.pmedr.2018.10.003. eCollection 2018 Dec. PMID 30406005
- [Background] Radesky JS, Christakis DA. Increased Screen Time: Implications for Early Childhood Development and Behavior. Pediatr Clin North Am. 2016 Oct;63(5):827-39. doi: 10.1016/j.pcl.2016.06.006. PMID 27565361
- [Background] Guideline: Sugars Intake for Adults and Children. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK285537/ PMID 25905159
- [Background] Roberts CA, Giesbrecht T, Fallon N, Thomas A, Mela DJ, Kirkham TC. A Systematic Review and Activation Likelihood Estimation Meta-Analysis of fMRI Studies on Sweet Taste in Humans. J Nutr. 2020 Jun 1;150(6):1619-1630. doi: 10.1093/jn/nxaa071. PMID 32271923
- [Background] van Loveren C. Sugar Restriction for Caries Prevention: Amount and Frequency. Which Is More Important? Caries Res. 2019;53(2):168-175. doi: 10.1159/000489571. Epub 2018 Aug 8. PMID 30089285
- [Background] Schulze MB, Manson JE, Ludwig DS, Colditz GA, Stampfer MJ, Willett WC, Hu FB. Sugar-sweetened beverages, weight gain, and incidence of type 2 diabetes in young and middle-aged women. JAMA. 2004 Aug 25;292(8):927-34. doi: 10.1001/jama.292.8.927. PMID 15328324
- [Background] Sim E, Sohn W, Choi ES, Noh H. Sugar-sweetened beverage consumption frequency in Korean adolescents: based on the 2015 Youth Risk Behavior Web-Based Survey. Int Dent J. 2019 Oct;69(5):376-382. doi: 10.1111/idj.12485. Epub 2019 May 11. PMID 31077367
- [Background] Moynihan P, Makino Y, Petersen PE, Ogawa H. Implications of WHO Guideline on Sugars for dental health professionals. Community Dent Oral Epidemiol. 2018 Feb;46(1):1-7. doi: 10.1111/cdoe.12353. Epub 2017 Nov 23. PMID 29168887
- [Background] Weinstein A, Livny A, Weizman A. New developments in brain research of internet and gaming disorder. Neurosci Biobehav Rev. 2017 Apr;75:314-330. doi: 10.1016/j.neubiorev.2017.01.040. Epub 2017 Feb 11. PMID 28193454
- [Background] Hale L, Guan S. Screen time and sleep among school-aged children and adolescents: a systematic literature review. Sleep Med Rev. 2015 Jun;21:50-8. doi: 10.1016/j.smrv.2014.07.007. Epub 2014 Aug 12. PMID 25193149
- [Background] Orgiles M, Owens J, Espada JP, Piqueras JA, Carballo JL. Spanish version of the Sleep Self-Report (SSR): factorial structure and psychometric properties. Child Care Health Dev. 2013 Mar;39(2):288-95. doi: 10.1111/j.1365-2214.2012.01389.x. Epub 2012 Jun 8. PMID 22676274
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Vereecken CA, Maes L. A Belgian study on the reliability and relative validity of the Health Behaviour in School-Aged Children food-frequency questionnaire. Public Health Nutr. 2003 Sep;6(6):581-8. doi: 10.1079/phn2003466. PMID 14690039
- [Background] Fisher JO, Serrano EL, Foster GD, Hart CN, Davey A, Bruton YP, Kilby L, Harnack L, Ruth KJ, Kachurak A, Lawman HG, Martin A, Polonsky HM. Title: efficacy of a food parenting intervention for mothers with low income to reduce preschooler's solid fat and added sugar intakes: a randomized controlled trial. Int J Behav Nutr Phys Act. 2019 Jan 17;16(1):6. doi: 10.1186/s12966-018-0764-3. PMID 30654818
- [Derived] Restrepo-Serna C, Caicedo-Giraldo M, Velasquez-Baena L, Bonfanti G, Santamaria-Villegas A. Effect of Screen Time and Sugar Consumption Reduction on Sleep Bruxism in Children: A Randomised Clinical Trial. J Oral Rehabil. 2025 Apr;52(4):506-520. doi: 10.1111/joor.13913. Epub 2025 Jan 9. PMID 39789814